CLINICAL TRIAL: NCT06744231
Title: Thriving Hearts: Healing-Centered, Integrated, Community Maternity Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Orange County Health Department (Unknown); Duke University (Other); Wake Forest University Health Sciences (Other); The North Carolina Alliance of Public Health Agencies, Inc. (Unknown); Jacaranda Health (Other); Piedmont Health Services, Inc. (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-2138
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Hypertensive Disorder of Pregnancy
Keywords: Community health workers; Medical Legal Partnership; Home blood pressure monitoring; Low dose aspirin; Community Resilience Model; Trauma-informed care; Healing Centered Engagement; Sense of community; Person-centered maternity care
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Intervention Model Description: The investigators plan a multisite step-wedge cluster randomized trial to test the extent to which the a Local Health Department led population health program reduces rates of hypertensive disorders of pregnancy (HDP, primary outcome), patient experience measures (secondary outcomes) and maternity health worker quality of life (secondary outcome). The Thriving Hearts program will be implemented in a stepped-wedge design with six nine-month time periods, 3 sequences, and 3 or 4 counties in each sequence, with 10 counties in total.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (Placebo Comparator): In the pre-intervention sequence(s), pregnant and parenting people in participating counties will experience treatment-as-usual.
  Interventions: Other: Usual Care
- Post-intervention (Active Comparator): In the post-intervention sequence(s), pregnant and parenting people in participating counties will experience care enhanced with Thriving Hearts components, including point-of-care HDP prevention, health care providers equipped with resources for coping with secondary trauma, and proactive provision of social and material support.
  Interventions: Behavioral: Thriving Hearts

INTERVENTIONS:
Other: Usual Care — Prior to implementation of the Thriving Hearts package of services, people living in participating counties will receive usual care for pregnancy, birth, and postpartum services. The study team will quantify existing services using a study-developed usual care assessment instrument.
  Arms: Pre-intervention
Behavioral: Thriving Hearts — Thriving Hearts is a collaboration among LHDs in ten North Carolina counties. At the individual level, pregnant individuals will self-screen for HDP risk during prenatal visits, and those at risk will be provided a Mama Hearts Care Kit, including a home blood pressure monitor, low dose aspirin, and culturally tailored educational materials.
  At the healthcare provider level, burnout and compassion fatigue will be addressed through skill-building activities, including training in the Community Resilience and Mindfulness-Based Stress Reduction.
  At the community level, Loving Connection will provide proactive material and social support through Community Health Workers, text messaging-based communication, a medical legal partnership, and capacity-building support for community-based organizations.
  Arms: Post-intervention

SUMMARY:
The overarching goal of Thriving Hearts is to implement a multi-level program through Local Health Departments (LHDs) that cultivates conditions for mothers and birthing people to not only survive pregnancy, but to thrive. Thriving Hearts is a collaboration among LHDs in ten North Carolina counties, designed to reduce incidence of Hypertensive Disorders of Pregnancy (HDP) and their complications through support and connection at the individual, healthcare provider, and community level. The investigators will conduct a pragmatic, stepped-wedge, cluster randomized study. Participating LHDs will begin in a usual care phase, and they will transition to Thriving Hearts in clusters in a randomly assigned sequence at 9-month intervals.

DETAILED DESCRIPTION:
Birthing people in the United States experience unacceptable rates of severe maternal morbidity (SMM) and maternal mortality (MM). Hypertensive disorders of pregnancy (HDP) are a major contributor: among individuals who died during the birth hospitalization, one in three had an HDP diagnosis. Populations that have experienced structural racism are disproportionately affected. Compared with white birthing people, Black birthing people with HDP are more likely to experience severe morbidity, and they are 3.7 times more likely to die from HDP complications. To address the root causes of these disparities, multicomponent strategies are urgently needed. The overarching goal of Thriving Hearts is to implement such a multi-level intervention through Local Health Departments (LHDs), cultivating conditions for mothers and birthing people to not only survive pregnancy, but to thrive. Thriving Hearts is a collaboration among LHDs in ten North Carolina counties, designed to reduce incidence of HDP and its complications through support and connection at the individual, healthcare provider, and community level. At the individual level, Mama Hearts maternity care will provide evidence-based, culturally tailored, holistic preventative care for pregnant people at risk for HDP. At the healthcare provider level, the project will address burnout and compassion fatigue among LHD staff and community healthcare providers through healing-centered, trauma-informed care. At the community level, Loving Connection will deploy community health workers and an integrated medical-legal partnership to provide proactive support through universal, strength-based assistance in a mutual aid context, building awareness of local resources and cultivating spaces for community support, connection, and joy.

The Thriving Hearts study uses a hybrid type 1 effectiveness-implementation design. To quantify effectiveness, the team will conduct a pragmatic, stepped-wedge, cluster randomized trial, implementing the intervention through LHDs. Participating LHDs will begin in a usual care phase, and they will transition to Thriving Hearts in pairs in a randomly assigned sequence, at 9-month intervals. The team will systematically document usual care in each county. To inform future scale-up and dissemination, the team will conduct a mixed methods implementation evaluation.

The team will use this approach to accomplish the following specific aims: 1) Quantify the extent to which Thriving Hearts reduces incidence of HDP and associated complications and increases uptake of support resources among birthing people in the ten Thriving Hearts counties, using PCORnet, Carolina Cost and Quality Initiative Claims, Birth Certificate, and State Hospital Discharge data. 2) Quantify the extent to which Thriving Hearts improves patient-reported experiences and outcomes, measured through cross-sectional surveys of a subset of postpartum people in each county. 3) Quantify the extent to which healing-centered, trauma-informed care improves health team effectiveness and well-being, measured using cross-sectional surveys of professional quality of life and wellbeing. 4) Identify factors that affect implementation of the Thriving Hearts program at health department- and community-levels using the Consolidated Framework for Implementation Research 2.0.

The study population will include all individuals who give birth in the 10 Thriving Hearts counties, including Alamance, Caswell, Chatham, Cumberland, Durham, Forsyth, Guilford, Johnston, Orange, and Person Counties. In 2021, there were 26,900 births in these counties, of whom 29% were non-Hispanic Black, 19% were Hispanic, and 43% were non-Hispanic white. Over the five-year comparative effectiveness study, the team anticipates that there will be ~140,000 births in the participating counties, providing ample power to assess outcomes in the full sample and to perform stratified analyses to test the extent to which Thriving Hearts reduces disparities in processes, experiences, and outcomes.

The study's primary outcome is the incidence of HDP during pregnancy, birth, or within 28 days postpartum, indexed by clinical data (PCORnet), diagnosis codes, and documentation on the birth certificate. Among Thriving Hearts county residents who birthed at UNC-affiliated hospitals from January 2019 through March 2023, 20.4% of Black patients and 17.4% of white patients had a diagnosis of HDP. The team hypothesizes that Thriving Hearts will reduce HDP incidence by 20%, consistent with effect sizes reported for several subcomponents of the multilevel intervention.

Secondary outcomes include clinical processes (first-trimester enrollment Medicaid and WIC, postpartum visit attendance, acute care utilization) and outcomes (HDP morbidity, severe maternal morbidity); patient-reported experiences (person-centered maternity care, autonomy, respectful care) and outcomes (wellbeing, mental health, social support, maternal function); and health care team-reported experience (addressing health-related social needs) and outcomes (wellbeing, professional quality of life, secondary trauma symptoms).

ELIGIBILITY:
Any individual who is pregnant or <4 months postpartum and resides in county where Thriving Hearts is active can engage with Thriving Hearts-supported programs and services.

Cross-sectional survey of postpartum people

For participation in the population-based survey of postpartum parents, the following criteria are required:

Inclusion Criteria:

* Age ≥15 and ≤55
* Had a live birth at >=24 weeks in the past 6 months
* Listed the birthing parent's residential address on the birth certificate as within a Thriving Hearts county ( Alamance, Caswell, Chatham, Cumberland, Durham, Forsyth, Guilford, Johnston, Orange, and Person counties)
* Are able to communicate in English or Spanish

Exclusion Criteria

* < 15 or > 55 years of age
* Did not have a live birth at >= 24 weeks in the past 6 months
* Residential address not listed on birth certificate as one of the study counties
* Not able to communicate in either English

Cross-sectional survey of people who serve perinatal patients

To assess the effectiveness of the Healing Centered Engagement program, the team will conduct cross-sectional surveys of people who serve perinatal patients in Thriving Hearts counties, repeated during each of the six study time periods

Inclusion criteria:

* Age ≥ 18
* Provides services for perinatal patients in a Thriving Hearts county (Alamance, Caswell, Chatham, Cumberland, Durham, Forsyth, Guilford, Johnston, Orange, and Person counties)
* Are able to communicate in English

Exclusion criteria:

* Age < 18
* Does not provide services for perinatal patients in a Thriving Hearts county (Alamance, Caswell, Chatham, Cumberland, Durham, Forsyth, Guilford, Johnston, Orange, and Person counties)
* Are unable to communicate in English

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17500 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Hypertensive Disorder of Pregnancy | Between admission for delivery and 4 weeks postpartum
  Population-level incidence of hypertensive disorders of pregnancy.

SECONDARY OUTCOMES:
Change in Brief Professional Quality of Life Score among people who serve pregnant women in Thriving Hearts Counties | Cross-sectional survey of individuals who serve pregnant women in Thriving Hearts counties, repeated during each of the six study time periods, at months 6, 15, 24, 33, 42, and 51.
  The Brief Professional Quality of Life scale is a measure of compassion satisfaction, burnout, and secondary traumatic stress. assessed using a 5-point Likert scale: 1 = Never (0 days), 2 = Rarely (1 day), 3 = Sometimes (2-3 days), 4 = Often (4-5 days), 5 = Always (6-7 days). Scores range from 12-60 with higher scores associated with worse professional quality of life.
Change in World Health Organization (WHO)-5 Wellbeing Index among people who serve pregnant women in Thriving Hearts Counties | Cross-sectional survey of individuals who serve pregnant women in Thriving Hearts counties, repeated during each of the six study time periods, at months 6, 15, 24, 33, 42, and 51.
  The WHO-5 is a short questionnaire consisting of 5 simple and non-invasive statements rated using Likert questions ranging from 5 (all the time) to 0 (never), which tap into the subjective well-being of the respondents. Scores range from 0-100 (raw score is multiplied by 4). Higher scores = higher wellbeing.
Person-Centered Maternity Care Scale Score, postpartum survey | Cross-sectional survey of postpartum people in Thriving Hearts counties 2-6 months following birth
  The Person-Centered Maternity Care Scale is a validated tool that can be used to measure person-centered prenatal care that reflects the experiences of people of color consisting of 26 items. Scores range from a minimum of 16 to a maximum of 78 with higher scores indicate more person-centered care.
Brief Sense of Community Scale, postpartum survey | Cross-sectional survey of postpartum people in Thriving Hearts counties 2-6 months following birth
  The BSCS was designed to assess the dimensions of needs fulfillment, group membership, influence, and emotional connection with 8 questions rated using a 5-point, Likert-type response option format ranging from strongly agree to strongly disagree. Scores range from 8-40 wtih higher scores indicating a stronger sense of community.
World Health Organization (WHO)-5 Wellbeing Index, postpartum survey | Cross-sectional survey of postpartum people in Thriving Hearts counties 2-6 months following birth
  The WHO-5 is a short questionnaire consisting of 5 simple and non-invasive statements rated using Likert questions ranging from 5 (all the time) to 0 (never), which tap into the subjective well-being of the respondents. Scores range from 0-100 (raw score is multiplied by 4). Higher scores = higher wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Stuebe, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 to 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- See also: PCORI: Thriving Hearts: Healing-Centered, Integrated, Community Maternity Care — https://www.pcori.org/research-results/2023/thriving-hearts-healing-centered-integrated-community-maternity-care